CLINICAL TRIAL: NCT02005575
Title: The Effect of Dexamethasone on the Duration and Functionality of Bupivacaine Intercostal Nerve Blockade
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, dermot Maher, Resident Department of Anesthesia, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00032069
Record Dates: First submitted 2013-11-05; First posted 2013-12-09 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Post Minimally Invasive Thorascopic Surgical Pain
MeSH Terms: interventions — Bupivacaine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Group 1 (Placebo Comparator): an intercostal nerve block with a solution consisting of 0.46% bupivicaine (19.5 ml of 0.5% bupivicaine + .5ml normal saline)
  Interventions: Drug: Placebo
- Group 2 (Active Comparator): an intercostal nerve block with a solution consisting of 0.46% bupivicaine (19.5 ml of 0.5% bupivicaine + .5ml .4% dexamethasone)
  Interventions: Drug: Bupivacaine and Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine and Dexamethasone — The standard of care is to use a regional block solution containing both decadron and bupivicaine.
  Other Names: Decadron
  Arms: Group 2
Drug: Placebo
  Arms: Group 1

SUMMARY:
The proposed study is a randomized, double-blinded, non-placebo-controlled evaluation of the effect of the addition of dexamethasone to intraoperative intercostal nerve block bupivicaine solutions on the duration of pain relief and post operative pulmonary function.

DETAILED DESCRIPTION:
Our study proposes two groups of 25 patients undergoing similar VATS surgery with a single surgeon, Dr. R. McKenna, who will receive interoperatively placed intercostal nerve blocks at the same levels. Each group will receive intercostals nerve blocks with one of two different solutions: group one will receive intercostal nerve blocks with only 0.46% bupivacaine (19.5 ml of 0.5% bupivacaine + .5 cc saline), group 2 will receive intercostal blocks with 0.46% bupivacaine and dexamethasone(19.5 ml of 0.5% bupivacaine + .5ml .4% dexamethasone). The patients will have pulmonary lung function objectively assessed by portable spirometry and clinical factors both preoperatively and postoperatively. Our study objective is to examine and quantify the potentially beneficial effects of intercostal nerve blockade prolongation with dexamethasone on postoperative pulmonary function and postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years old of either gender, scheduled for unilateral VATS procedure with Dr. McKenna for resection of lung tumor.

Exclusion Criteria:

* ASA IV and above
* Intolerance, allergy, or contraindication to use of any medications used in this study
* Significant coronary artery disease (abnormal stress test, myocardial infarction within the last 3 months)
* Uncontrolled hypertension (BP > 140/90)
* History of prior ipsilateral thorascopic surgery
* Cardiac arrhythmias particularly prolonged QT syndrome
* Drugs known to cause prolonged qT: class IA antiarrhythmics (quinidine, procainamide, dysopyramide), class III antiarrhythmics (sotalol, dofetalide, ibutalide, amiodarone), haloperidol, thioridazine, arsenic trioxide, HIV protease inhibitors, tricyclic antidepressants
* Individuals with significant psychological disorders including: schizophrenia, mania, bipolar disorder or psychosis
* Pregnant or lactating women
* Morbid obesity (BMI > 40 kg/m2) AND/OR weight > 150 kg
* Chronic renal failure ( creatinine > 2.0 mg/dL)
* Liver failure e.g., active cirrhosis
* Alcohol or substance abuse within in the past 3 months
* Uncorrected hypokalemia, hypomagnesemia, hypocalcemia (can be due to diuretics, mineralocorticoid use, laxatives)
* Restrictive lung disease (pulmonary fibrosis, myasthenia gravis) or FEV1 or FEV less than 70% of predicted value.
* Type 2 diabetes
* Neuropathic pain
* Chronic opioid consumption (>30mg oxycodone or greater per day)
* Cahexia from any cause
* systemic use of corticosteroids for greater than 2 weeks in the 6 months prior to surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 72 hours post operatively
  Patients will be evaluated for post operative pain using the NRS pain evaulation

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States